CLINICAL TRIAL: NCT02281591
Title: Disposition of Eslicarbazepine Acetate and Its Metabolites S-licarbazepine and R-licarbazepine Following Oral Administration in Healthy Volunteers
Brief Title: Disposition of Eslicarbazepine Acetate and Its Metabolites S-licarbazepine and R-licarbazepine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BIA-2093-115
Record Dates: First submitted 2014-10-30; First posted 2014-11-03 (Estimated); Results first posted 2014-12-03 (Estimated); Last update posted 2025-04-08 (Actual); Status verified 2025-03

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy | interventions — eslicarbazepine acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- eslicarbazepine acetate (Experimental): 900mg of eslicarbazepine acetate (ESL, BIA 2-093)
  Interventions: Drug: BIA 2-093
- S-licarbazepine R-licarbazepine (Active Comparator): 450 mg of S-licarbazepine plus 450 mg of R-licarbazepine
  Interventions: Drug: S-licarbazepine; Drug: R-licarbazepine
- S-licarbazepine (Active Comparator): 450 mg of S-licarbazepine
  Interventions: Drug: S-licarbazepine
- R-licarbazepine (Active Comparator): 450 mg of Rlicarbazepine
  Interventions: Drug: R-licarbazepine

INTERVENTIONS:
Drug: BIA 2-093 — Tablets containing 900 mg
  Arms: eslicarbazepine acetate
Drug: S-licarbazepine — capsules containing 225 mg
  Arms: S-licarbazepine; S-licarbazepine R-licarbazepine
Drug: R-licarbazepine — capsules containing 225 mg
  Arms: R-licarbazepine; S-licarbazepine R-licarbazepine

SUMMARY:
Single centre, open-label, randomised study in four parallel groups of healthy volunteers

DETAILED DESCRIPTION:
Single centre, open-label, randomised study in four parallel groups of healthy volunteers: Group 1 = 900 mg of eslicarbazepine acetate (ESL, BIA 2-093); Group 2 = 450 mg of S-licarbazepine plus 450 mg of R-licarbazepine; Group 3 = 450 mg of S-licarbazepine; Group 4 = 450 mg of Rlicarbazepine. In each group, the study consisted of a single-dose period (Phase A) followed by a repeateddose period of 7 days of duration in which the investigational product was administered once daily (Phase B). The repeated-dose phase started 96 h post single-dose.

ELIGIBILITY:
Inclusion Criteria

* Male or female subjects aged between 18 and 45 years, inclusive.
* Subjects of body mass index (BMI) between 19 and 30 kg/m2, inclusive.
* Subjects who were healthy as determined by pre-study medical history, physical examination, vital signs, neurological examination, and 12-lead ECG.
* Subjects who had clinical laboratory tests clinically acceptable at screening and admission.
* Subjects who had negative tests for HBsAg, anti-HCV Ab and HIV-1 and HIV-2 Ab at screening.
* Subjects who were negative for drugs of abuse and alcohol at screening and admission.
* Subjects who were non-smokers or who smoke < 10 cigarettes or equivalent per day.
* Subjects who are able and willing to give written informed consent.
* (If female) She was not of childbearing potential by reason of surgery or, if of childbearing potential, she used one of the following methods of contraception: double barrier, intrauterine device or abstinence.
* (If female) She had a negative pregnancy test at screening and admission to Phase A.

Exclusion Criteria:

* Subjects who did not conform to the above inclusion criteria, OR
* Subjects who had a clinically relevant history or presence of respiratory, gastrointestinal, renal, hepatic, haematological, lymphatic, neurological, cardiovascular, psychiatric, musculoskeletal, genitourinary, immunological, dermatological, endocrine, connective tissue diseases or disorders.
* Subjects who had a clinically relevant surgical history.
* Subjects who had a clinically relevant family history.
* Subjects who had a history of relevant atopy.
* Subjects who had a history of relevant drug hypersensitivity (especially carbamazepine or oxcarbazepine).
* Subjects who had a history of alcoholism or drug abuse.
* Subjects who consumed more than 14 units of alcohol a week.
* Subjects who had a significant infection or known inflammatory process on screening or admission.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2006-06; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Scope International Life Sciences AG,, Hamburg, Germany

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Eslicarbazepine Acetate | S-licarbazepine R-licarbazepine | S-licarbazepine | R-licarbazepine
Started | 8 | 8 | 8 | 8
Completed | 8 | 8 | 8 | 8
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Eslicarbazepine Acetate | S-licarbazepine R-licarbazepine | S-licarbazepine | R-licarbazepine | Total
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 8 | 8 | 8 | 32
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 4 | 4 | 16
  Male | 4 | 4 | 4 | 4 | 16

OUTCOME MEASURES:

1. Primary Outcome: Cmax - the Maximum Plasma Concentration
Description: BIA 2-194, BIA 2-195 and Oxcarbazepine are metabolites of BIA 2-093 and Licarbazepine.
Time Frame: Phase A: pre-dose (Day 1); and ½, 1, 1½, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72 and 96 hours post-dose.Phase B: Days 6 to 10 inclusively: pre-dose. Day 11 (last dose): pre-dose; and ½, 1, 1½,2, 3, 4, 6, 8, 12, 16, 24, 36, 48, 72 and 96 hours post-dose.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Eslicarbazepine Acetate | S-licarbazepine R-licarbazepine | S-licarbazepine | R-licarbazepine
Number analyzed (Participants) | 8 | 8 | 8 | 8
ng/mL
  Cmax (BIA 2-194) | 15809 (3183) | 10496 (1432) | 10364 (3352) | 437 (143)
  Cmax (BIA 2-195) | 222 (68.4) | 8099 (1258) | 132 (29.6) | 6941 (1054)
  Cmax (Oxcarbazepine) | 136 (25.1) | 261 (53.5) | 92.8 (21.8) | 101 (28.6)

2. Primary Outcome: Tmax - the Time of Occurrence of Cmax
Description: BIA 2-194, BIA 2-195 and Oxcarbazepine are metabolites of BIA 2-093 and Licarbazepine.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Eslicarbazepine Acetate | S-licarbazepine R-licarbazepine | S-licarbazepine | R-licarbazepine
Number analyzed (Participants) | 8 | 8 | 8 | 8
hours
  tmax (BIA 2-194) | 1.99 (0.916) | 1.01 (0.320) | 0.965 (0.496) | 10.7 (3.69)
  tmax (BIA 2-195) | 18.6 (4.14) | 1.41 (0.320) | 11.7 (3.77) | 1.22 (0.582)
  tmax (Oxcarbazepine) | 3.59 (1.61) | 1.34 (0.354) | 1.36 (1.44) | 1.21 (0.641)

3. Primary Outcome: AUC0-∞ - the Area Under the Plasma Concentration Versus Time Curve From Time Zero to Infinity
Description: BIA 2-194, BIA 2-195 and Oxcarbazepine are metabolites of BIA 2-093 and Licarbazepine.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng.h/mL
Arm/Group | Eslicarbazepine Acetate | S-licarbazepine R-licarbazepine | S-licarbazepine | R-licarbazepine
Number analyzed (Participants) | 8 | 8 | 8 | 8
ng.h/mL
  AUC0-∞ (BIA 2-194) | 271191 (47416) | 201409 (37377) | 132724 (20175) | 11003 (4476)
  AUC0-∞ (BIA 2-195) | 8816 (2168) | 116884 (22425) | 5417 (824) | 66087 (16072)
  AUC0-∞ (Oxcarbazepine) | 3181 (1078) | 4726 (1163) | 2500 (1923) | 1073 (793)

4. Secondary Outcome: AUC0-t - the Area Under the Plasma Concentration-time Curve to Last Measurable Time Point
Description: BIA 2-194, BIA 2-195 and Oxcarbazepine are metabolites of BIA 2-093 and Licarbazepine.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng.h/mL
Arm/Group | Eslicarbazepine Acetate | S-licarbazepine R-licarbazepine | S-licarbazepine | R-licarbazepine
Number analyzed (Participants) | 8 | 8 | 8 | 8
ng.h/mL
  AUC0-t (BIA 2-194) | 268045 (46861) | 198313 (38771) | 130147 (19326) | 9419 (4707)
  AUC0-t (BIA 2-195) | 6757 (2211) | 114635 (21741) | 3074 (1001) | 65203 (16161)
  AUC0-t (Oxcarbazepine) | 1947 (757) | 3401 (902) | 748 (308) | 422 (247)

ADVERSE EVENTS:
Arm/Group | Eslicarbazepine Acetate | S-licarbazepine R-licarbazepine | S-licarbazepine | R-licarbazepine
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 6/8 | 8/8 | 4/8 | 5/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Eslicarbazepine Acetate (N=8) | S-licarbazepine R-licarbazepine (N=8) | S-licarbazepine (N=8) | R-licarbazepine (N=8)
Burning sensation in eye (Eye disorders) | 1 | 0 | 0 | 0
Visual disturbance (Eye disorders) | 0 | 0 | 0 | 1
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Numbness of tongue (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Oral dryness (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Paraesthesia lips (Gastrointestinal disorders) | 0 | 2 | 1 | 0
Paraesthesia tongue (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Feeling hungry (General disorders) | 1 | 0 | 0 | 0
Tiredness (General disorders) | 1 | 6 | 1 | 2
Vaginal infection (Infections and infestations) | 0 | 0 | 0 | 1
Accidental injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Leg pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Acroparaesthesia (Nervous system disorders) | 1 | 0 | 0 | 0
Concentration loss (Nervous system disorders) | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 0 | 0 | 0
Head pressure (Nervous system disorders) | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 3 | 3 | 1 | 1
Increased libido (Psychiatric disorders) | 0 | 0 | 0 | 1
Blister of fingers, without mention of infection (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Herpes labialis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Itching (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Bulla dorsum manus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Tooth extraction (Surgical and medical procedures) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other